CLINICAL TRIAL: NCT04372667
Title: Adaptation and Evaluation of the PMTCT Community Score Card Approach in Dedza and Ntcheu Districts, Malawi
Brief Title: Adaptation and Evaluation of the PMTCT CSC in Dedza and Ntcheu Districts, Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: Cooperative for Assistance and Relief Everywhere, Inc. (CARE) (Unknown); Centers for Disease Control and Prevention (U.S. Federal Agency); Ministry of Health, Malawi (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: EG0163
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: HIV/AIDS; Infant Morbidity
Keywords: PMTCT; HIV; Quality improvement; Social accountability; Patient centered; Retention in care; Early infant diagnosis of HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Community score card approach
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post intervention (Experimental): Community score card approach
  Interventions: Behavioral: Community score card approach

INTERVENTIONS:
Behavioral: Community score card approach — The CSC intervention is a participatory community approach. Health care workers (HCWs), PMTCT clients identified the issues that most impacted PMTCT service quality and uptake, and came together to implement actions for improvement. The core implementation strategy is using dialogue in a participatory forum that engages both service users and service providers. The CSC consists of five core phases, repeated on a regular basis (called "rounds"), for the life of the project. The five core phases include:
  1. Phase I: Planning and preparation
  2. Phase II: Conducting the Score Card with the community
  3. Phase III: Conducting the Score Card with service providers
  4. Phase IV: Interface meeting and action planning
  5. Phase V: Action plan implementation and follow-up
  Other Names: social accountability; user involvement; patient engagement

SUMMARY:
This CDC-funded study sought to evaluate the effect of an adapted Community Score Card Approach on maternal retention in ART, maternal retention across the PMTCT service cascade, and the uptake of early infant diagnosis services in Malawi. The study also estimated the cost of the implementation of the Community Score Card Approach.

DETAILED DESCRIPTION:
Prevention of Mother to Child HIV Transmission (PMTCT) services aim to identify HIV-infected pregnant and breastfeeding mothers and initiate them on antiretroviral treatment (ART) for improving the health of the mother as well as reducing HIV transmission to their infants. In 2011, Malawi was the first country to adopt lifelong ART for HIV- pregnant and breastfeeding women, known as 'Option B+'. Despite leading the way on operationalization of this approach, Malawi has faced challenges retaining HIV-infected pregnant and breastfeeding women on lifelong ART as well as with improving uptake of early infant HIV testing for HIV-exposed infants. Innovative approaches are needed which engage health service users (i.e. patients) as part of quality improvement solutions within clinical settings to improve retention throughout the PMTCT cascade and ultimately improve PMTCT outcomes for mothers and infants.

One approach to broadly engage health service users in quality improvement activities is the Community Score Card (CSC). The CSC engages both service providers and users within a clinical setting in dialogues to identify solutions to the perceived barriers with health service delivery and utilization.

CARE developed the CSC intervention in Malawi in 2002 as part of a project aimed at developing innovative and sustainable models to improve general maternal and child health services. The main goal of the CSC intervention is to positively influence the quality, efficiency, and accountability with which health services are provided at different levels. The original CSC consists of five core phases, repeated on a regular basis (called "rounds"), for the life of the project.

This project adapted the CSC to the PMTCT setting across 11 sites in two priority PEPFAR scale-up districts in Malawi. The adaptation of the CSC was evaluated through a pre-post design to measure change in maternal retention on ART, change in maternal retention across the PMTCT service cascade, and uptake of Early Infant Diagnosis (EID) services following CSC implementation. Additionally, the project estimated the cost of the adapted CSC implementation.

ELIGIBILITY:
Inclusion Criteria:

* New born infants of HIV-positive women
* Women 18 years and over newly initiating antiretroviral therapy (ART) at ART clinic
* HIV-positive pregnant women >15 years of age newly receiving care at first ANC (ANC1)
* Women who are HIV-positive at ANC1 (known positive, already on treatment)
* Women who are newly identified HIV-positive and initiated on treatment at ANC (newly identified at ANC or labor and delivery)
* Women known HIV-positive but not yet on treatment prior to enrollment at ANC and initiated on treatment at ANC

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1233 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Early diagnosis of HIV exposed infants (HEI) | 6 - 8 weeks after birth
  Proportion of HEI receiving a DNA PCR test
Early retention of pregnant and breastfeeding HIV positive women in PMTCT | 1 to 6 months
  Proportions of HIV-positive pregnant and breastfeeding women (including women newly-identified and already-known to be HIV positive) retained in PMTCT services
Early retention of newly diagnosed HIV-positive women in HIV care | 1 to 6 months
  Proportions of HIV-positive women (pregnant and breastfeeding women as well as non-pregnant women) newly initiating ART services retained in HIV care
Implementation cost of CSC | 12 months
  Estimate the total cost of implementing of the CSC intervention at community and facility levels.

CONTACTS AND LOCATIONS:
Overall Officials: Godfrey Woelk, PhD, Principal Investigator — E. Glaser Pediatric AIDS Found
Locations (1):
- Elizabeth Glaser Pediatric AIDS Foundation, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laterra A, Callahan T, Msiska T, Woelk G, Chowdhary P, Gullo S, Mwale PM, Modi S, Chauwa F, Kayira D, Kalua T, Wako E. Bringing women's voices to PMTCT CARE: adapting CARE's Community Score Card(c) to engage women living with HIV to build quality health systems in Malawi. BMC Health Serv Res. 2020 Jul 22;20(1):679. doi: 10.1186/s12913-020-05538-2. PMID 32698814